CLINICAL TRIAL: NCT03020420
Title: Clinical Trial To Study The Anti-scarring Effect Of Cicatricell
Acronym: Cicatricell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cicatricell
Record Dates: First submitted 2015-09-16; First posted 2017-01-13 (Estimated); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Surgical Incisions
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment arm (Experimental): receive cicatricell cream
  Interventions: Other: Cicatricell Cream
- control arm (No Intervention): to treatment

INTERVENTIONS:
Other: Cicatricell Cream — Cream to be applied 2 times a day for 8weeks to 6 months
  Arms: treatment arm

SUMMARY:
This study tries to prove that Cicatricell cream significantly reduces scarring with better wound appearance as compared to no treatment.

DETAILED DESCRIPTION:
At 1st post operative follow up visit, surgical incision(s) will be assessed for healing, after the sutures/staples/steri-strips are removed. To be included in the study the incision must be 5cm or greater. And bilateral incisions as in bilateral mastectomy can be included. The incisions will be divided into two sections, using an imaginary line between top and bottom, or left and right. One side of the imaginary line will have cicatricell cream applied 2 times a day for a minimum of 8 weeks and a maximum 6months. The other side of the imaginary line will remain untreated. In the case of a bilateral incision, as in bilateral breast mastectomy or AAA incisions in the groins, the cream will be applied to one entire incision and the 2nd incision will be untreated. The incision(s) will be its own control group. At the end of the treatment phase the incision(s) will be assessed again to compare the healing.

ELIGIBILITY:
Inclusion Criteria:

* Signed IRB approved, written informed consent.
* Patient from 18 to 60 years of age.
* Patient who recently underwent a surgery involving linear surgical skin incisions of 5cm or more or patients with two exactly symmetrical separate incisions like bilateral inguinal hernia repair or bilateral mastectomy, CT surgery patients will be included.

Exclusion Criteria:

* Known skin allergies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2015-03; Primary Completion 2018-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Improved wound appearance | 8 weeks to 6 months
  improved wound appearance by surface area measurement
improved wound appearance | 8 weeks to 6 months
  wound indentation measurement with caliper
improved wound appearance | 8 weeks to 6 months
  wound bulge measured with caliper
Modified Vancouver Scar Scale | 8 weeks to 6 months
  a scale of visual assessment of a scar
Manchester Scar Scale | 8 weeks to 6 months
  A new quantitative scale for clinical scar assessment

CONTACTS AND LOCATIONS:
Locations (1):
- UTMC, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No